CLINICAL TRIAL: NCT04493645
Title: Optimizing Clinical Outcomes for Patients With Chronic Ankle Instability Using Foot Intensive Rehabilitation
Brief Title: Ankle Instability Using Foot Intensive Rehabilitation
Acronym: FIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Hoch (Other)
Collaborators: University of Virginia (Other); Naval Health Research Center (U.S. Federal Agency); Marine Corps Base Camp Pendleton (Other)
Responsible Party: Sponsor-Investigator, Matthew Hoch, Associate Professor, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 58500; CDMRP-OR190060 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-07-20; First posted 2020-07-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-01

CONDITIONS: Ankle Injuries; Ankle Sprains
Keywords: chronic ankle instability; rehabilitation; injury
MeSH Terms: conditions — Ankle Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The investigators will compare clinical and innovative outcome measures collected at five time points between cohorts of patients with CAI that receive a standard of care (SOC) rehabilitation program compared to an innovative foot intensive rehabilitation (FIRE) program to determine if FIRE can further reduce the rate of re-injury, improve sensorimotor function, and reduce self-reported disability during the 24 months following the intervention.
Who Masked: Outcomes Assessor
Masking Description: The investigators collecting the outcomes will be blinded to group allocation. Separate investigators will be used for intervention delivery and outcomes assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Participants will be randomized to receive standard of care rehabilitation (SOC) for a period of 6 weeks.The investigators will prospectively follow participants assigned to the SOC group for 24 months following completion of their assigned SOC intervention.
  Interventions: Behavioral: Standard of Care Rehabilitation (SOC)
- Foot Intensive Rehabilitation (FIRE) (Experimental): Participants will be randomized to receive foot intensive rehabilitation (FIRE) for a period of 6 weeks.The investigators will prospectively follow participants assigned to the FIRE group for 24 months following completion of their assigned SOC intervention.
  Interventions: Behavioral: Foot Intensive Rehabilitation (FIRE)

INTERVENTIONS:
Behavioral: Standard of Care Rehabilitation (SOC) — 6 weeks of standard of care rehabilitation will be given designed to restore ankle joint range of motion, strength, postural control, and functional movement. Each participant will be expected to complete 2 supervised sessions and 3 unsupervised at home sessions per week.
  Arms: Standard of Care (SOC)
Behavioral: Foot Intensive Rehabilitation (FIRE) — 6 weeks of FIRE will be given along with elements of SOC. Each participant will be expected to complete 2 supervised sessions and 3 unsupervised at home sessions per week.
  Arms: Foot Intensive Rehabilitation (FIRE)

SUMMARY:
The overall objective of this study is to examine the effects of a 6-week foot-intensive rehabilitation (FIRE) program on lateral ankle sprain (LAS) re-injury rates, CAI symptoms, sensorimotor function, and self-reported disability in CAI patients.

DETAILED DESCRIPTION:
Lateral ankle sprains are one of the most common injuries sustained by the general population with the greatest rates in people who are physically active or service members. Approximately 40% of lateral ankle sprain patients develop chronic ankle instability (CAI) characterized by recurrent lateral ankle sprains, repetitive sensations of ankle "giving way", residual ankle sprain symptoms, and self-reported disability. Factors related to the development and progression of CAI has been thoroughly studied. However, few interventions have been developed which have successfully created long term reductions in re-injury rates, physical function, or health-related quality of life. Recent work by our research team has uncovered several novel motor and sensory deficits in the foot in patients with CAI. Deficits in foot function may contribute to the high re-injury rates, deficits in balance and strength, and diminished health-related quality of life commonly experienced by individuals with CAI. The investigators expect the additive effect of FIRE with components of the standard of care (balance training, strength training, and range of motion) will create the synergy needed to reduce future injuries (Aim 1), enhance physical function (Aim 2), and reduce self-reported disability in CAI patients (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-44.
2. Previous history of at least 1 ankle sprain and at least 2 episodes of "giving way" in the past 3 months.
3. Participants must answer "yes" to at least 5 questions on the Ankle Instability Instrument.
4. Score of 11 or higher on the Identification of Functional Ankle Instability (IdFAI).
5. Confirmed clinical presentation of CAI by a PT, AT, or MD.

Exclusion Criteria:

1. Sustained an ankle sprain in the previous four weeks or lower extremity neuromusculoskeletal injury other than to the ankle in the last 12 months.
2. History of surgery to the lower extremity.
3. Sustained a lower extremity fracture.
4. History of neurological disease, vestibular or visual disturbance or any other pathology that would impair their sensorimotor performance.
5. Current participation in a formal ankle joint rehabilitation program.
6. Sustained a concussion in the last 12 months.
7. Exhibit clinical examination characteristics of foot and ankle function which are consistent with conditions other than CAI (i.e. fracture, deformity).

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of recurrent ankle sprains | 24 months
  The ability of FIRE to attenuate the occurrence of ankle sprains compared to SOC rehabilitation will be determined through self-report. An ankle sprain will be operationally defined as an incident in which the rearfoot was inverted or supinated and resulted in a combination of swelling, pain, and time lost or modification of normal function for at least one day.
Frequency of episodes of the ankle giving way | 24 months
  The ability of FIRE to attenuate the number of episodes of the ankle giving way compared to SOC rehabilitation will be determined through self-reported occurrences per week in the past month. Episodes of giving way will be operationally defined for the subject as an incident in which the rearfoot suddenly rolled, felt weak, or lost stability; however, the individual did not sustain an ankle sprain and was able to continue with normal function.
Severity of chronic ankle instability related symptoms | 24 months
  The ability of FIRE to attenuate the severity of related symptoms compared to SOC rehabilitation will be determined through the Cumberland Ankle Instability Tool. The Cumberland Ankle Instability Tool is a 9-item instrument used to identify self-reported impairments associated with CAI. This instrument is scored on a 0-30 scale, where lower scores represent greater severity of CAI related symptoms.

SECONDARY OUTCOMES:
Postural Control | 24 months
  The ability of FIRE to improve static and dynamic postural control compared to SOC rehabilitation will be determined. Multiple measurements will be made including: Single-limb stance on each limb with eyes open and eyes closed with use of a force plate for center of pressure measurements, Star Excursion Balance Test, forward jump single limb landing stabilization task. All measurements will be monitored while the participant wears an inertial sensor placed on the lumbar spine.
Ankle/Toe Strength | 24 months
  The ability of FIRE to improve strength compared to SOC rehabilitation will be determined. Strength of the muscles surrounding the ankle and the toes will be assessed through a series of assessments with a digital handheld dynamometer.
Intrinsic Foot Muscle Activation | 24 months
  The ability of FIRE to improve foot muscle activation compared to SOC rehabilitation will be determined. Abductor hallucis, flexor digitorum brevis, quadratus plantae, and flexor hallucis brevis functional activity ratios will be captured using diagnostic ultrasound with a 12-4 MHz linear array transducer probe and measured using Image J software.
Plantar Cutaneous Sensation | 24 months
  The ability of FIRE to improve plantar cutaneous sensation compared to SOC rehabilitation will be determined. Plantar cutaneous sensation will be tested using a 20-piece Semmes-Weinstein Monofilament kit which has monofilaments ranging from to 0.008g of force (1.65 level) to 300g of force (6.65 level). Light touch detection thresholds will be assessed on the plantar surface at the 1st metatarsal head.

OTHER OUTCOMES:
Self-Reported Ankle Function | 24 months
  The ability of FIRE to improve disability outcomes compared to SOC rehabilitation will be determined. Self-reported disability will be assessed using the Foot and Ankle Ability Measure (FAAM). Sports and activities of daily living subscale scores will be calculated.
Self-Reported Disability | 24 months
  The ability of FIRE to improve disability outcomes compared to SOC rehabilitation will be determined. Self-reported disability will be assessed using the Disablement in the Physically Active Scale (DPA).
Self-Reported Fear Avoidance Beliefs | 24 months
  The ability of FIRE to improve disability outcomes compared to SOC rehabilitation will be determined. Self-reported disability will be assessed using the Fear Avoidance Beliefs Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hoch, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoch MC, Hertel J, Gribble PA, Heebner NR, Hoch JM, Kosik KB, Long D, Sessoms PH, Silder A, Torp DM, Thompson KL, Fraser JJ. Effects of foot intensive rehabilitation (FIRE) on clinical outcomes for patients with chronic ankle instability: a randomized controlled trial protocol. BMC Sports Sci Med Rehabil. 2023 Apr 9;15(1):54. doi: 10.1186/s13102-023-00667-7. PMID 37032355